CLINICAL TRIAL: NCT02441205
Title: The Impact of High Intensity Interval Training on Inflammatory State and Immune Function in Elderly Individuals
Brief Title: Interval Training, Inflammation and Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00055208
Record Dates: First submitted 2015-04-09; First posted 2015-05-12 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-02

CONDITIONS: Aging; Disease
Keywords: High Intensity Interval Training
MeSH Terms: conditions — Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIIT Aging (Experimental): all subjects will undergo high intensity interval training 3 x per week for 10-12 weeks. the intervals of high-intensity (~85% of maximal capacity) will be 5 to 10 bouts of 30 seconds at this intensity with rest periods in between intervals that range from 30 seconds to 2 minutes
  Interventions: Behavioral: High Intensity Interval training

INTERVENTIONS:
Behavioral: High Intensity Interval training — all subjects will undergo high intensity interval training 3 x per week for 10-12 weeks. the intervals of high-intensity (~85% of maximal capacity) will be 5 to 10 bouts of 30 seconds at this intensity with rest periods in between intervals that range from 30 seconds to 2 minutes

SUMMARY:
PURPOSE: The purpose of this study is to investigate whether High Intensity Interval Training (HIIT)can improve the health and wellbeing of pre-diabetic elderly adults. In particular, there is specific interest in describing the effects of an interval exercise program on inflammatory state and immune function.

DESIGN: Subjects will be sedentary, 65 to 80 years old adults, with prediabetes as defined by fasting plasma glucose (100 to 125 mg/dl). Before and after a 10-12 week High Intensity Interval Exercise training program subjects will undergo several tests including: 1) a maximal treadmill test, 2) an Oral Glucose Tolerance Test, 3) muscle biopsy, 4) body composition, 5) several physical function tests and 6) other health related measures including lung function, arterial stiffness and several blood measures (e.g. liver enzymes, kidney function).

DATA ANALYSES & SAFETY ISSUES: As there are no comparison groups, data analyses will consist of performing paired t-tests on pre and post exercise training values for each of the measurement variables of interest. In addition, the data will be used to provide power calculations for future grant proposals. High Intensity Interval Training is a very safe exercise modality. The regular use of vigorous intensity exercise intervals have been used extensively in exercise training. In fact, the exercise intervals will start at levels lower and will be of shorter duration than were used during the maximal exercise test. They will then be carefully and slowly made to be more challenging as each subject is able to safely tolerate.

HYPOTHESIS: The investigators hypothesize that HIIT will result in significant improvements in markers of inflammation, immune system markers and other health-related risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-80 years
* Prediabetic - Fasting plasma glucose is 100 - 125 on two separate days
* Able to walk for 2 minutes or more without stopping
* LDL Cholesterol ≤ 190; Triglycerides < 600;
* Blood Pressure ≤ 160/90
* Inactive: Exercise < 2 days per week
* Medications: Stable use of all medications ≥ three months

Exclusion Criteria:

* Smoker: tobacco use within the last 12 months
* Dieting or intending to diet; not weight stable ≥ six months (weight change < 5 pounds)
* Use of confounding inflammatory medications: aspirin, ibuprofen, naproxen (NSAIDS - nonsteriodal anti-inflammatory drugs)
* History of diabetes, heart disease or taking medications for those conditions
* History of hypertension (high blood pressure) not controlled with medication
* Unwillingness to undergo muscle biopsies and all other study testing, or to continuously participate in exercise training for 12 weeks.
* Inability to give blood continuously through a catheter (please notify the study nurse of any difficulties you have had in the past when having your blood drawn; the study nurse will determine whether you are excluded for this reason)
* Unwillingness to conduct ALL exercise sessions at the fitness facility during research study staff supervised times.
* Orthopedic limitations, musculoskeletal disease and/or injury Due to the nature of the study, persons with known joint, muscle or other orthopedic limitations that restrict physical activity may be excluded.
* Able to decide if you want to take part in the study
* Lack of transportation to the exercise and testing facilities

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory markers in plasma | baseline and following exercise training, approximately 10-12 weeks
Change in inflammatory markers in muscle | baseline and following exercise training, approximately 10-12 weeks
Change in immune markers in peripheral blood | baseline and following exercise training, approximately 10-12 weeks
Change in immune markers in muscle | baseline and following exercise training, approximately 10-12 weeks

SECONDARY OUTCOMES:
Change in Metabolic Syndrome risk factors composite score | baseline and following exercise training, approximately 10-12 weeks
  Classic and additional Metabolic Syndrome measures include: blood pressure, waist circumference, triglycerides, HDL, fasting glucose; plus liver and kidney function, insulin sensitivity, glucose tolerance, etc...

OTHER OUTCOMES:
Change in Physical Function outcome measures composite score | baseline and following exercise training, approximately 10-12 weeks
  Peak VO2, 400 meter walk time, short physical performance battery (SPPB)

CONTACTS AND LOCATIONS:
Overall Officials: William Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

REFERENCES:
- [Derived] Bartlett DB, Slentz CA, Willis LH, Hoselton A, Huebner JL, Kraus VB, Moss J, Muehlbauer MJ, Spielmann G, Muoio DM, Koves TR, Wu H, Huffman KM, Lord JM, Kraus WE. Rejuvenation of Neutrophil Functions in Association With Reduced Diabetes Risk Following Ten Weeks of Low-Volume High Intensity Interval Walking in Older Adults With Prediabetes - A Pilot Study. Front Immunol. 2020 May 5;11:729. doi: 10.3389/fimmu.2020.00729. eCollection 2020. PMID 32431698